CLINICAL TRIAL: NCT01125371
Title: Computerized BI for Binge Drinking HIV At-Risk and Infected African-American Women
Brief Title: Computerized Brief Alcohol Intervention (BI) for Binge Drinking HIV At-Risk and Infected Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAAGC018632; R01AA018632 (NIH)
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Results first posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Alcohol; Harmful Use; Binge Drinking; Risk Behavior; HIV Infection
Keywords: Hazardous alcohol use; Binge drinking; High risk sexual behaviors; HIV risk reduction
MeSH Terms: conditions — Binge Drinking; Risk-Taking; HIV Infections | interventions — Ethanol; Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Computerized Brief Alcohol Intervention + IVR (Experimental): Computer-delivered brief alcohol intervention (CBI) with booster phone calls delivered by IVR+ text messages (TM)
  Interventions: Behavioral: Computerized brief alcohol intervention + IVR booster calls
- Computerized Brief Alcohol Intervention (Active Comparator): Computerized Brief Alcohol Intervention only (CBI)
  Interventions: Behavioral: Computerized brief alcohol intervention
- Attention Control (Placebo Comparator): Attention control
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Computerized brief alcohol intervention + IVR booster calls — 1) Computerized brief alcohol intervention + IVR booster calls: Clinic-based computerized brief alcohol intervention (delivered once) followed by three booster phone calls using interactive voice response technology + text messages
  Other Names: CBI+IVR+TM
  Arms: Computerized Brief Alcohol Intervention + IVR
Behavioral: Computerized brief alcohol intervention — Computerized brief alcohol intervention: Clinic based computer delivered brief alcohol intervention delivered one time
  Other Names: CBI
  Arms: Computerized Brief Alcohol Intervention
Behavioral: Attention Control — Attention Control: 20 minute attention control condition focused on dental hygiene delivered once
  Arms: Attention Control

SUMMARY:
African American (AA) women are disproportionately affected by HIV/AIDs. The major risk factor for HIV acquisition among AA women is high-risk heterosexual sex, including unprotected vaginal and anal sex, and sex with a high-risk partner. Hazardous alcohol use has been associated with high risk sexual behaviors and prevalent gonorrhea among women attending an urban STI clinic, both of which increase a woman's vulnerability to HIV acquisition and transmission. This application proposes a randomized controlled trial (RCT) of a culturally tailored computer-directed brief alcohol intervention (CBI) enhanced with cell-phone booster calls using interactive voice response technology (IVR) and text messages among HIV-infected and at-risk AA women attending an urban STI Clinic. Hazardous drinking AA women (N=450) presenting with STI complaints will be randomized to one of three arms: 1) usual clinical care, 2) clinic-based, CBI, or 3) clinic-based, CBI + 3 booster calls using IVR and text messages. The CBI, an evidence-based based method for behavior change, will use principles of motivational interviewing, to counsel on: 1) alcohol use and 2) associated HIV/STI risk behaviors. Primary outcomes, measured at 3, 6, and 12 month intervals, include alcohol-related risk behaviors (number of binge drinking episodes, drinking days/week, and drinks per occasion), sexual risk behaviors (number of partners, episodes of unprotected vaginal/anal sex, episodes of sex while high), and occurrence of HIV/STI biomarkers. Prior to implementing the RCT, the CBI and IVR software messages will be revised to: 1) include the association between hazardous alcohol use and risky sexual behaviors, and 2) ensure their relevance and acceptability using quantitative/qualitative feedback from a sample of AA women attending a Baltimore City STI clinic. The proposed research focuses on a particularly vulnerable population of urban HIV at-risk and HIV-infected AA women seeking treatment in a public STI clinic and examines two novel BI intervention delivery strategies specifically tailored to be culturally/socially relevant to this minority population. If the intervention(s) prove to be effective, study findings will offer "real life" specialty care clinics a screening and intervention package that is practical, low cost, and easy to implement.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. HIV infected or HIV negative and attending the Baltimore City Health Department sexually transmitted infection clinic for STI-related services
3. Consumes an average of 8 or more drinks per week OR has had two binge drinking episodes (4 drinks/occasion) in the last 3 months
4. sexually active
5. Cognitively able to understand proposed research design (10 min screening, followed by random assignment to one of three study groups (if individual fulfills criteria for RCT enrollment);
6. Able to speak and understand English
7. Able and willing to receive text messages

Exclusion Criteria:

1. Pregnant women will be excluded and referred directly to social work for referral to either alcohol or drug treatment due to ethical concerns of randomization to usual care.
2. Currently enrolled in alcohol or drug treatment.
3. Non-English Speaking.
4. Actively Psychotic or have other severe mental health symptoms that would prevent appropriate participation in the brief intervention protocol.
5. Planning on moving out of the area within 12 months of study entry

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2011-10; Primary Completion 2016-06-07 (Actual); Study Completion 2016-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geetanjali Chander, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Baltimore City Health Department STD Clinic, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Computerized Brief Alcohol Intervention + IVR | Computerized Brief Alcohol Intervention | Attention Control
Started | 146 | 145 | 148
3 Months Follow up | 127 | 131 | 135
6 Months Follow up | 125 | 133 | 131
12 Months Follow up | 120 | 130 | 129
Completed | 120 | 130 | 129
Not Completed | 26 | 15 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Computerized Brief Alcohol Intervention + IVR | Computerized Brief Alcohol Intervention | Attention Control | Total
Number analyzed (Participants) | 146 | 145 | 148 | 439
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [25 to 43] | 31 [25 to 45] | 31 [24 to 45] | 31 [25 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 145 | 148 | 439
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 131 | 125 | 132 | 388
  Other | 15 | 20 | 16 | 51
Level of Education [Count of Participants; unit: Participants]
  < Grade 12 | 42 | 41 | 50 | 133
  GED or Higher | 104 | 104 | 98 | 306
Income [Count of Participants; unit: Participants]
  $0 - 5,000 | 77 | 63 | 75 | 215
  $5,001 - 10,000 | 23 | 35 | 25 | 83
  $10,001 - 15,000 | 18 | 24 | 22 | 64
  $15,001 or more | 28 | 23 | 26 | 77
HIV Positive Status [Count of Participants; unit: Participants]
  No | 132 | 129 | 140 | 401
  Yes | 8 | 10 | 4 | 22
  Unsure | 6 | 6 | 4 | 16
Illicit Drug Use [Count of Participants; unit: Participants] | 95 | 93 | 97 | 285
Marijuana Use [Count of Participants; unit: Participants] | 78 | 72 | 71 | 221
Cocaine Use [Count of Participants; unit: Participants] | 21 | 21 | 20 | 62
Heroin Use [Count of Participants; unit: Participants] | 16 | 9 | 7 | 32
Injection Drug Use [Count of Participants; unit: Participants] | 3 | 2 | 1 | 6
Non-medical Use of Prescription [Count of Participants; unit: Participants] | 9 | 16 | 12 | 37
PHQ Depressive Symptoms [Median (Inter-Quartile Range); unit: score on a scale] — Patient Health Questionnaire (PHQ) assesses for depressive symptoms: The score range is 0-27. Diagnosis Total Score For Score Action Minimal depression 0-4, Mild depression 5-9, Moderate depression 10-14, Moderately severe depression 15-19, Severe depression 20-27.
  score on a scale | 6 [3 to 10] | 7 [3 to 12] | 7.5 [4 to 12] | 7 [3 to 11]
PHQ Panic Symptoms [Count of Participants; unit: Participants] — Participants with Panic Symptoms per the PHQ assessment.
  Participants | 35 | 52 | 43 | 130
Post-Traumatic Stress Disorder (PTSD) [Count of Participants; unit: Participants] — Participants with Post-Traumatic Stress Disorder.
  Participants | 46 | 51 | 54 | 151
Generalized Anxiety Symptoms [Count of Participants; unit: Participants]
  None | 81 | 63 | 72 | 216
  Mild | 39 | 45 | 43 | 127
  Moderate | 15 | 20 | 20 | 55
  Severe | 10 | 17 | 13 | 40
  Missing | 1 | 0 | 0 | 1
MINI Assessment [Count of Participants; unit: Participants] — The MINI Assessment is an assessment for alcohol abuse or dependence. It assesses for the Diagnostic and Statistical Manual of Mental Disorders (DSM) Alcohol use Disorder, categorized as "Neither", "Abuse" or "Dependence".
  Participants
    Neither | 54 | 42 | 45 | 141
    Abuse | 23 | 32 | 26 | 81
    Dependence | 69 | 71 | 77 | 217
Audit Score [Count of Participants; unit: Participants] — The Audit Score is an Alcohol use disorders identification test which assesses alcohol use. Scores range from 0-40.
  <7 = no hazardous alcohol use
  7-12 = Hazardous alcohol use
  ≥13 = Alcohol use Disorder
  Participants
    <7 | 40 | 35 | 43 | 118
    7-12 | 34 | 47 | 47 | 128
    ≥13 | 72 | 63 | 58 | 193

OUTCOME MEASURES:

1. Primary Outcome: Change in Alcohol Use (Heavy Drinking Days)
Description: Change in alcohol-related risk behavior as assessed by the number of heavy drinking days.
Time Frame: Baseline, 3, 6, and 12 months
Population: Some participants in each of the arms did not complete assessments at 3, 6 and 12 months.
Measure: Median (Inter-Quartile Range); unit: heavy drinking days
Arm/Group | Computerized Brief Alcohol Intervention + IVR | Computerized Brief Alcohol Intervention | Attention Control
Number analyzed (Participants) | 146 | 145 | 148
heavy drinking days
  Baseline | 6 [2 to 13] | 6 [3 to 11] | 6 [2 to 11]
  3 months: number analyzed (Participants) | 125 | 130 | 135
  3 months | 3 [1 to 7] | 3 [1 to 8] | 3 [0 to 8]
  6 months: number analyzed (Participants) | 125 | 133 | 131
  6 months | 3 [0 to 7] | 4 [1 to 8] | 2 [0 to 8]
  12 months: number analyzed (Participants) | 119 | 130 | 129
  12 months | 2 [0 to 6] | 2 [0 to 6] | 3 [1 to 6]

2. Primary Outcome: Change in Alcohol Use (Drinking Days)
Description: Change in alcohol-related risk behavior as assessed by the number of drinking days.
Time Frame: Baseline, 3, 6, and 12 months
Population: Some participants in each of the arms did not complete assessments at 3, 6 and 12 months.
Measure: Median (Inter-Quartile Range); unit: drinking days
Arm/Group | Computerized Brief Alcohol Intervention + IVR | Computerized Brief Alcohol Intervention | Attention Control
Number analyzed (Participants) | 146 | 145 | 148
drinking days
  Baseline | 9 [5 to 15] | 9 [6 to 14] | 8.5 [5.8 to 15]
  3 months: number analyzed (Participants) | 125 | 130 | 135
  3 months | 6.4 [3 to 10] | 7 [4 to 12] | 6 [2.1 to 11]
  6 months: number analyzed (Participants) | 125 | 133 | 131
  6 months | 6 [2 to 11] | 7 [2 to 12] | 5 [2 to 11]
  12 months: number analyzed (Participants) | 119 | 130 | 129
  12 months | 6 [2 to 11] | 6 [2 to 11] | 6 [2 to 10]

3. Primary Outcome: Change in Alcohol Use (Drinks Per Drinking Day)
Description: Change in alcohol-related risk behavior as assessed by the standard drinks per drinking day.
Time Frame: Baseline, 3, 6, and 12 months
Population: Some participants in each of the arms did not complete assessments at 3, 6 and 12 months.
Measure: Median (Inter-Quartile Range); unit: drinks per drinking day
Arm/Group | Computerized Brief Alcohol Intervention + IVR | Computerized Brief Alcohol Intervention | Attention Control
Number analyzed (Participants) | 146 | 145 | 148
drinks per drinking day
  Baseline | 5.6 [3.2 to 8.8] | 5.6 [3.3 to 9.3] | 6.1 [3.7 to 7.8]
  3 months: number analyzed (Participants) | 125 | 130 | 135
  3 months | 3.7 [2.2 to 6.2] | 4.2 [2.3 to 6.4] | 4.1 [2.0 to 6.5]
  6 months: number analyzed (Participants) | 125 | 133 | 131
  6 months | 3.8 [1.4 to 6.4] | 4.4 [2.1 to 6.8] | 3.8 [1.7 to 6.2]
  12 months: number analyzed (Participants) | 119 | 130 | 129
  12 months | 3.0 [1.5 to 5.7] | 3.4 [1.4 to 5.6] | 3.8 [1.4 to 6.5]

4. Primary Outcome: Change in Alcohol Use (Drinks Per Week)
Description: Change in alcohol-related risk behavior as assessed by the standard drinks per week.
Time Frame: Baseline, 3, 6, and 12 months
Population: Some participants in each of the arms did not complete assessments at 3, 6 and 12 months.
Measure: Median (Inter-Quartile Range); unit: drinks per week
Arm/Group | Computerized Brief Alcohol Intervention + IVR | Computerized Brief Alcohol Intervention | Attention Control
Number analyzed (Participants) | 146 | 145 | 148
drinks per week
  Baseline | 12.0 [4.7 to 28.7] | 12.4 [5.8 to 25.5] | 12.0 [5.3 to 25.3]
  3 months: number analyzed (Participants) | 125 | 130 | 135
  3 months | 6.5 [2.1 to 13.6] | 7.0 [2.9 to 15.4] | 6.4 [1.6 to 16.1]
  6 months: number analyzed (Participants) | 125 | 133 | 131
  6 months | 5.6 [1.1 to 13.1] | 6.8 [1.4 to 15.7] | 4.4 [0.9 to 15.7]
  12 months: number analyzed (Participants) | 119 | 130 | 129
  12 months | 4.3 [1.0 to 11.5] | 5.3 [1.0 to 12.4] | 5.4 [1.4 to 11.2]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Computerized Brief Alcohol Intervention + IVR | Computerized Brief Alcohol Intervention | Attention Control
All-Cause Mortality (participants affected / at risk) | 1/146 | 0/145 | 1/148
Serious Adverse Events (participants affected / at risk) | 0/146 | 0/145 | 0/148
Other Adverse Events (participants affected / at risk) | 0/146 | 0/145 | 0/148

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT01125371/Prot_SAP_000.pdf